CLINICAL TRIAL: NCT01364389
Title: A 2-week Single-blind, Randomized, 3-arm Proof of Concept Study of the Effects of AIN457 (Anti-IL17 Antibody), ACZ885 (Canakinumab, Anti-IL1b Antibody), or Corticosteroids in Patients With Polymyalgia Rheumatica, Followed by an Open Label Phase to Assess Safety and Long Term Efficacy
Brief Title: A 3-arm Proof of Concept Study of AIN457, ACZ885 or Corticosteroids in Patients With Polymyalgia Rheumatica
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data did not show that the two biologic treatments impacted PMR disease activity to the same degree as steroid treatment within a 2-week treatment period.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPJMR0012201; 2010-019395-73 (EudraCT Number)
Record Dates: First submitted 2011-03-10; First posted 2011-06-02 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Polymyalgia Rheumatica; Inflammatory Diseases
Keywords: Polymyalgia Rheumatica; Inflammatory Disease; Rheumatic Disease
MeSH Terms: conditions — Polymyalgia Rheumatica; Rheumatic Diseases | interventions — secukinumab; canakinumab; Prednisone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- ACZ885 (Experimental): On day 1, patients received a single intravenous dose of ACZ885 3mg/kg along with a placebo intravenous infusion in a double dummy manner to maintain the blind. On day 15, partial and complete responders continued in the open label phase of this treatment arm where they were eligible to receive one re-dose of ACZ885 upon confirmed disease flare. Non-responders started a 20 mg dose cycle of prednisone or prednisolone followed by standard steroid tapering.
  Interventions: Drug: AIN457; Drug: Placebo
- AIN457 (Experimental): On day 1, patients received a single intravenous dose of AIN457 3mg/kg along with a placebo intravenous infusion in a double dummy manner to maintain the blind. On day 15, partial and complete responders continued in the open label phase of this treatment arm where they were eligible to receive one re-dose of AIN457 upon confirmed disease flare. Non-responders started a 20 mg dose cycle of prednisone or prednisolone followed by standard steroid tapering.
  Interventions: Drug: ACZ885; Drug: Placebo
- Prednisone (Other): On day 1, patients received daily oral doses of prednisone 20 mg along with daily oral placebo doses to in a double-dummy manner to maintain the blind. On day 15, partial and complete responders continued in the study and tapered their steroid treatment according to standard care. Non-responders were discontinued from the study.
  Interventions: Drug: Prednisone; Drug: Placebo

INTERVENTIONS:
Drug: AIN457 — 3 mg/kg
  Arms: ACZ885
Drug: ACZ885 — 3 mg/kg
  Other Names: canakinumab
  Arms: AIN457
Drug: Prednisone — 20 mg
  Arms: Prednisone
Drug: Placebo — Matching placebo to AIN457, ACZ885 and prednisone

SUMMARY:
The study is a two-week, single-blinded, double-dummy, randomized, active-controlled, parallel group design, with a follow-up period up to a total study duration of 6-month, non-randomized, open-label phase to monitor safety, tolerability and, in responders, flare. It is a multicentric, multinational study. The protocol will seek to enroll a total of 30 patients, who will be randomized to the 3 arms at a ratio of 1:1:1.

Patients will have a maximum screening period of 7 days with randomization at D1 for a dosing period of 15 days followed by a follow up-period of 154 days, or 4 months (112 days) after their last biologic dose, whichever is greater, and followed by unblinded re-dosing in the case of a disease flare.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following features:
* Patients ≥ 50 and ≤ 85 years
* C-reactive protein (CRP) > 1.0 mg/dl OR erythrocyte sedimentation rate (ESR) > 30 mm/hr
* New bilateral shoulder and/or hip pain
* Early morning stiffness ≥ 60 min
* Duration of illness > 1 week
* A negative 5 U purified protein derivative skin test (PPD) skin test (≤ 5 mm induration) at screening

Exclusion Criteria:

* Active infection or current use of antibiotics
* Known human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatits B virus (HBV)
* Previous therapy with methotrexate or other immunosuppressive agents within three months prior to baseline
* History of malignancy other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix within five years prior to study entry
* Presence of rheumatoid arthritis or other inflammatory arthritic processes (features of Giant Cell Artertitis (GCA), spondyloarthropathies), connective tissue disease, drug-induced myopathies, endocrine disorders, neurological disorders, chronic pain syndromes, as assessed by base line screening including thyroid-stimulating hormone (TSH), creatine kinase (CK), rheumatoid factor (RF), cyclic citrullinated peptide (CCP), antinuclear antibodies (ANA), serum protein electrophoresis, urinalysis.

Other protocol-defined inclusion/exclusion criteria apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-02-14 (Actual); Primary Completion 2013-01-29 (Actual); Study Completion 2013-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Novartis Investigative Site, Rochester, Minnesota, United States
- Novartis Investigative Site, Berlin, Germany
- Italy (2):
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Siena, SI
- United Kingdom (2):
  - Novartis Investigative Site, Basildon, Essex
  - Novartis Investigative Site, Westcliff-on-Sea, Essex

REFERENCES:
- [Derived] Sun MM, Pope JE. Polymyalgia rheumatica and giant cell arteritis: diagnosis and management. Curr Opin Rheumatol. 2025 Jan 1;37(1):32-38. doi: 10.1097/BOR.0000000000001059. Epub 2024 Oct 14. PMID 39400109

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACZ885 | AIN457 | Prednisone
Started | 5 | 6 | 5
Pharmacodynamic (PD) Analysis Set | 5 | 6 | 4 (One patient excluded: did not receive study drug; received placebo caps. and infusion only in error.)
Completed | 3 | 5 | 4
Not Completed | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Protocol deviation | 0 | 0 | 1
Not completed — Administrative problems | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACZ885 | AIN457 | Prednisone | Total
Number analyzed (Participants) | 5 | 6 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (9.09) | 68.8 (8.61) | 69.4 (7.89) | 68.5 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 11
  Male | 1 | 4 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Polymyalgia Rheumatica Activity Score (PMR-AS)
Description: The efficacy of a single dose of AIN457 and ACZ885 (canakinumab) was measured by the polymyalgia rheumatica activity score. A composite PMR-AS was developed from the following components: measure of C-reactive protein (CRP), measure of Erythrocyte Sedimentation Rate (ESR), assessment of early morning stiffness, assessment of the patient's elevation on upper limbs, patient's assessment of pain, and physician's global assessment of disease activity. Treatment effect was measured by the percent reduction in PMR-AS. N=3 for the ACZ885 arm because CRP values at Day 15 were missing for 2 participants.
Time Frame: Baseline, Day 15
Population: Pharmacodynamic (PD) Analysis Set: This set included participants who received at least one dose of study medication and had no major protocol deviation that may impact the PD data.
Measure: Least Squares Mean (Standard Error); unit: Percent reduction
Arm/Group | ACZ885 | AIN457 | Prednisone
Number analyzed (Participants) | 3 | 6 | 4
Percent reduction | 64.5 (0.68) | 51.7 (0.47) | 91.9 (86.2)

2. Secondary Outcome: Time to Partial Clinical Response
Description: The time to partial clinical response was assessed in patients who received a single dose of AIN457 or ACZ885 (canakinumab). Daily monitoring (home-based) of CRP was performed. This outcome shows the percentage of patients who achieved a partial clinical response at Day 15. A participant was defined as a partial responder if the participant had:
  >50% reduction in patient global assessment visual analogue scale (VAS) compared with baseline and morning stiffness < 60 minutes.
Time Frame: Day 15
Population: PD analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | ACZ885 | AIN457 | Prednisone
Number analyzed (Participants) | 5 | 6 | 4
Percentage of participants | 20.0 | 16.7 | 75.0

3. Secondary Outcome: Time to Complete Clinical Response
Description: The time to complete clinical response was assessed in patients who received a single dose of AIN457 or ACZ885 (canakinumab). Daily monitoring (home-based) of CRP was performed. This outcome shows the percentage of patients who achieved a complete clinical response at Day 15. A participant was defined as a complete responder if the participant had: >70% reduction in patient global assessment VAS compared with baseline, morning stiffness < 30 min, CRP < 1.0 mg/dL and/or ESR < 30 mm/1st hr.
Time Frame: Day 15
Population: PD analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | ACZ885 | AIN457 | Prednisone
Number analyzed (Participants) | 5 | 6 | 4
Percentage of participants | 0.0 | 0.0 | 25.0

4. Secondary Outcome: Time to First Flare
Description: This study was terminated because the data did not show that the two biologic treatments impacted PMR disease activity to the same degree as steroid treatment within a 2-week treatment period. Only 1 participant experienced a flare, in the AIN457 treatment group. The flare for this one participant occurred on study day 44
Time Frame: 6 months
Population: This study was terminated because the data did not show that the two biologic treatments impacted PMR disease activity to the same degree as steroid treatment within a 2-week treatment period. Only 1 participant experienced a flare, in the AIN457 treatment group. The flare for this one participant occurred on study day 44
Measure: Number; unit: Days
Arm/Group | ACZ885 | AIN457 | Prednisone
Number analyzed (Participants) | 0 | 1 | 0
Days |  | 44 |

5. Secondary Outcome: Number of Flares Over a 6 Month Period
Description: This study was terminated because the data did not show that the two biologic treatments impacted PMR disease activity to the same degree as steroid treatment within a 2-week treatment period. The summary statistics include patients with a valid measurements for the outcome measure.
Time Frame: 6 months
Population: This study was terminated because the data did not show that the two biologic treatments impacted PMR disease activity to the same degree as steroid treatment within a 2-week treatment period. The summary statistics include patients with a valid measurements for the outcome measure.
Measure: Number; unit: Participant
Arm/Group | ACZ885 | AIN457 | Prednisone
Number analyzed (Participants) | 0 | 1 | 0
Participant |  | 1 |

6. Secondary Outcome: Mean Steroid Dose Over a 6 Month Period
Description: as for outcome 5
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Number of doses
Arm/Group | ACZ885 | AIN457 | Prednisone
Number analyzed (Participants) | 3 | 4 | 4
Number of doses | 276.8 (46.34) | 256.7 (27.89) | 428.9 (131.44)

7. Secondary Outcome: Number of Patients Who Experienced Adverse Events, Serious Adverse Events and Deaths
Time Frame: 6 months
Population: Safety analysis set: This set included all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | ACZ885 | AIN457 | Prednisone
Number analyzed (Participants) | 5 | 6 | 5
Participants
  Adverse Events (serious and non-serious) | 3 | 2 | 5
  Serious Adverse Events | 0 | 0 | 0
  Deaths | 0 | 0 | 0

8. Secondary Outcome: Comparison Between the Initial Response to AIN457 and ACZ885 and the Response After Re-dosing of AIN457 and ACZ885 - Assessed by the Number of Flares After Redosing.
Description: One participant experienced one flare after initial dose but this participant had no flare after a redose. This patient was in the AIN457 arm.
Time Frame: 6 months
Population: One participant experienced one flare after initial dose but this participant had no flare after a redose. This patient was in the AIN457 arm.
Arm/Group | ACZ885 | AIN457 | Prednisone
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Effect on Health-related Quality of Life Via the Short Form-36 (SF-36) Questionnaire
Description: The Short Form-36 (SF-36) Questionnaire is a 36-item questionnaire yields an 8-scale health profile as well as summary measures of individual patients.. The scores range for each subscale from 0 to 10, and the composite score ranges from 0 to 100, with higher scores indicative of better health.
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ACZ885 | AIN457 | Prednisone
Number analyzed (Participants) | 5 | 6 | 4
Scores on a scale
  Physical component score at baseline | 26.126 (8.1517) | 29.009 (4.3115) | 27.001 (5.2561)
  Physical component score at EOS / Month 6 (n=4,6,2): number analyzed (Participants) | 4 | 6 | 2
  Physical component score at EOS / Month 6 (n=4,6,2) | 44.293 (12.6038) | 48.496 (8.2306) | 34.544 (7.7632)
  Mental component score at baseline | 30.490 (11.2875) | 35.779 (5.9113) | 29.673 (6.1925)
  Mental component score at month 6 / EOS (n=4,6,2): number analyzed (Participants) | 4 | 6 | 2
  Mental component score at month 6 / EOS (n=4,6,2) | 44.668 (20.3716) | 54.136 (8.8815) | 55.233 (2.8274)

10. Secondary Outcome: Effect on Health-related Quality of Life Via the Health Assessment Questionnaire (HAQ)
Description: HAQ: The scores range from 0 (min) to 3 (max). Higher scores = more disability; lower scores = less disability.
Time Frame: baseline and at month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ACZ885 | AIN457 | Prednisone
Number analyzed (Participants) | 5 | 6 | 4
Scores on a scale
  standard disability score at baseline | 1.900 (0.6869) | 1.646 (0.2896) | 2.063 (0.2394)
  standard disability score at EOS / Month 6 (n=4,6,3): number analyzed (Participants) | 4 | 6 | 3
  standard disability score at EOS / Month 6 (n=4,6,3) | 0.719 (1.0225) | 0.188 (0.3513) | 0.958 (0.3819)

11. Secondary Outcome: Effect on Health-related Quality of Life Via the Health Assessment Questionnaire (HAQ) - % Change From Baseline in the Standard Disability Score at EOS / Month 6
Description: HAQ: The scores range from 0 (min) to 3 (max). Higher scores = more disability; lower scores = less disability.
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | ACZ885 | AIN457 | Prednisone
Number analyzed (Participants) | 4 | 6 | 3
Percentage | -68.06 (36.781) | -86.83 (25.478) | -54.04 (12.296)

12. Secondary Outcome: Pharmacokinetics of AIN457 and ACZ885 - Cmax
Time Frame: Day 15
Population: This study was terminated because the data did not show that the two biologic treatments impacted PMR disease activity to the same degree as steroid treatment within a 2-week treatment period. The summary statistics include patients with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: microgram/mL
Arm/Group | ACZ885 | AIN457
Number analyzed (Participants) | 4 | 3
microgram/mL | 69.9 (5.58) | 46.8 (2.85)

13. Secondary Outcome: Pharmacokinetics of AIN457 and ACZ885 - Tmax
Time Frame: Day 15
Population: as for outcome 12
Measure: Median (Full Range); unit: days
Arm/Group | ACZ885 | AIN457
Number analyzed (Participants) | 4 | 3
days | 0.0868 [0.0833 to 1.97] | 0.107 [0.0868 to 0.167]

14. Secondary Outcome: Pharmacokinetics of AIN457 and ACZ885 - AUCinf and AUClast
Time Frame: Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: microg/day/mL
Arm/Group | ACZ885 | AIN457
Number analyzed (Participants) | 3 | 2
microg/day/mL
  AUCinf (microg/day/mL) | 1570 (80) | 1260 (134)
  AUClast (microg/day/mL) | 1560 (74.7) | 1200 (132)

15. Secondary Outcome: Pharmacokinetics of AIN457 and ACZ885 - CL
Time Frame: Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | ACZ885 | AIN457
Number analyzed (Participants) | 3 | 2
L/day | 0.171 (0.440) | 0.157 (0.0106)

16. Secondary Outcome: Pharmacokinetics of AIN457 and ACZ885 - Vz
Time Frame: Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L
Arm/Group | ACZ885 | AIN457
Number analyzed (Participants) | 3 | 2
L | 6.49 (1.19) | 9.85 (1.29)

17. Secondary Outcome: Pharmacokinetics of AIN457 and ACZ885 - T1/2
Time Frame: Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | ACZ885 | AIN457
Number analyzed (Participants) | 3 | 4
Day | 26.6 (2.38) | 40.2 (4.47)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 239 days
Groups:
- ACZ885 3mg/kg: On day 1, patients received a single intravenous dose of ACZ885 3mg/kg along with a placebo intravenous infusion in a double dummy manner to maintain the blind. On day 15, partial and complete responders continued in the open label phase of this treatment arm where they were eligible to receive one re-dose of ACZ885 upon confirmed disease flare. Non-responders started a 20 mg dose cycle of prednisone or prednisolone followed by standard steroid tapering.
- AIN457 3mg/kg: On day 1, patients received a single intravenous dose of AIN457 3mg/kg along with a placebo intravenous infusion in a double dummy manner to maintain the blind. On day 15, partial and complete responders continued in the open label phase of this treatment arm where they were eligible to receive one re-dose of AIN457 upon confirmed disease flare. Non-responders started a 20 mg dose cycle of prednisone or prednisolone followed by standard steroid tapering.
- Prednisone 20mg: On day 1, patients received daily oral doses of prednisone 20 mg along with daily oral placebo doses to in a double-dummy manner to maintain the blind. On day 15, partial and complete responders continued in the study and tapered their steroid treatment according to standard care. Non-responders were discontinued from the study.
Arm/Group | ACZ885 3mg/kg | AIN457 3mg/kg | Prednisone 20mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 2/6 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 3mg/kg (N=5) | AIN457 3mg/kg (N=6) | Prednisone 20mg (N=5)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was terminated because the data did not show that the two biologic treatments impacted PMR disease activity to the same degree as steroid treatment within a 2-week treatment period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.